CLINICAL TRIAL: NCT00367822
Title: Transdermal Lisuride: a Double-blind, Randomized, Active- and Placebo-controlled Multi-centre Phase III Efficacy Trial for the Treatment of Patients With Restless Legs Syndrome (RLS)
Brief Title: Transdermal Lisuride: a Trial for the Treatment of Patients With Restless Legs Syndrome (RLS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axxonis Pharma AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tulir 03/01; EudraCT No.: 2005-003549-16
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2010-01

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome; dopamine agonist; lisuride; ropinirole
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Lisuride; ropinirole

INTERVENTIONS:
Drug: Lisuride
Drug: Ropinirole
Drug: Placebo

SUMMARY:
The objective of this trial is to compare an individually optimized dose of the lisuride TTS patch against placebo and against an individually optimized dose of oral ropinirole (active- and placebo-controlled design) in idiopathic and uremic RLS patients with regard to efficacy, safety, and quality of life.

DETAILED DESCRIPTION:
Approximately 300 patients will be randomized to receive either lisuride, ropinirole or placebo in a 2:1:1 fashion. After completion of 12 weeks of double-blind treatment, eligible patients will have the option to continue treatment with the lisuride patch for further 36 weeks in an open-label extension of the study.

Primary outcome: Changes in the total score of the International Restless Legs Severity Scale (IRLS) from baseline to end of double-blind treatment (12 weeks) will be used as primary efficacy outcome measure.

Secondary objectives are to evaluate quality of life, safety and tolerability. After the double-blind period, long-term efficacy of lisuride will be assessed for further 36 weeks in an open-label extension of the study.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic or uremic RLS
* RLS Diagnostic Index (RLS-DI) > 10
* Total score in the IRLS Rating Scale ≥ 15 at baseline
* No previous treatment for RLS or insufficient current therapy

Exclusion Criteria:

* Secondary RLS, e.g. due to iron deficiency (exception: uremia)
* History or presence of sleep disorders other than RLS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300

PRIMARY OUTCOMES:
International Restless Legs Severity Scale (IRLS)

SECONDARY OUTCOMES:
RLS-6 scales
CGI

CONTACTS AND LOCATIONS:
Overall Officials: Heike Benes, MD, Principal Investigator — Somnibene GmbH
Locations (1):
- IMEREM GmbH, Nuremberg, Germany